CLINICAL TRIAL: NCT04022291
Title: A Randomised, Double-blind, Two-period Crossover, Euglycaemic Glucose Clamp Study in Healthy Volunteers to Demonstrate Pharmacokinetic and Pharmacodynamic Similarity of Biocon Insulin 70/30 and Humulin® 70/30
Brief Title: Comparison of Pharmacokinetic (PK) and Pharmacodynamic(PD) of Biocon Insulin 70/30 and Humulin® 70/30
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocon Limited (Industry)
Collaborators: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: EQ7030
Record Dates: First submitted 2019-07-04; First posted 2019-07-17 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Biocon Insulin 70/30 (Experimental): 0.4 IU/kg Dose per administration, Subcutaneous Route of administration
  Interventions: Biological: Biocon Insulin 70/30
- Humulin® 70/30 (Active Comparator): 0.4 IU/kg Dose per administration, Subcutaneous Route of administration
  Interventions: Biological: Humulin ®70/30

INTERVENTIONS:
Biological: Humulin ®70/30 — Humulin® 70/30 is a premixed suspension of human insulin of recombinant deoxyribonucleic acid (rDNA)origin, which contains 30% short-acting human soluble insulin and 70% intermediate-acting isophane insulin.
  Human insulin is produced by recombinant deoxyribonucleic acid (rDNA), technology utilizing a non-pathogenic laboratory strain of Escherichia coli.
  Arms: Humulin® 70/30
Biological: Biocon Insulin 70/30 — Biocon Insulin 70/30 is a premixed suspension of human insulin of recombinant deoxyribonucleic acid (rDNA)origin, which contains 30% short-acting human soluble insulin and 70% intermediate-acting isophane insulin.
  Biocon insulin is produced by recombinant deoxyribonucleic acid (rDNA) technology utilizing a non-pathogenic laboratory strain of Escherichia coli.
  Arms: Biocon Insulin 70/30

SUMMARY:
Two-centre, randomised, double-blind, single dose, two-treatment, two-period, two sequence, crossover, 24-hour euglycaemic glucose clamp trial in healthy subjects.

DETAILED DESCRIPTION:
The present study is designed to demonstrate pharmacokinetic and pharmacodynamic equivalence of Biocon Insulin 70/30 with Humulin® 70/30 in healthy subjects The treatment consists of one single dose of the test or reference product, administered during each of the two study periods, separated by 5-7 days between dosing. The planned trial duration for each subject is about 12 to 36 days.

Eligible subjects will undergo two 24-hour euglycaemic clamp examinations, one after administration of the test product and one after administration of the reference product in random order.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or post-menopausal female subjects. Post-menopausal state is defined as no menses for 12 months without an alternative medical cause and confirmed by a follicle stimulating hormone (FSH) level in the post-menopausal range (>= 25.8 IU/L).
* Age between 18 and 55 years, both inclusive.
* Body Mass Index (BMI) between 18.5 and 29.0 kg/m^2, both inclusive.
* Fasting plasma glucose concentration <= 100 mg/dL.
* Considered generally healthy upon completion of medical history and screening safety assessments, as judged by the Investigator.

Exclusion Criteria:

* Known or suspected hypersensitivity to Investigational Medicinal products ((IMP(s)) or related products.
* Receipt of any medicinal product in clinical development within 30 days or five times its half-life (whichever is longer) before randomization in this trial.
* Any history or presence of clinically relevant comorbidity, as judged by the investigator.
* Systolic blood pressure < 95 mmHg or >140 mmHg and/or diastolic blood pressure < 50 mm Hg or > 90 mmHg after resting for at least 5 minutes in supine position (excluding white-coat hypertension; therefore, a repeat test showing results within range will be acceptable).
* Pulse rate at rest outside the range of 50-90 beats per minute.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic endpoints: area under the insulin concentration curve (AUCins) 0-24h | 0-24hour
  area under the insulin concentration curve
Pharmacokinetic endpoints: insulin concentration (Cins).max | 0-24hour
  maximum observed insulin concentration.
Pharmacodynamic Endpoint: Area under curve (AUC)Glucose infusion rate (GIR).0-24h | 0-24hour
  area under the glucose infusion rate curve
Pharmacodynamic Endpoint: maximum glucose infusion rate (GIRmax) | 0-24hour
  maximum glucose infusion rate

SECONDARY OUTCOMES:
Pharmacokinetic endpoint: area under the insulin concentration curve(AUCins) 0-2h | 0-2hour
  area under the insulin concentration curve
Pharmacokinetic endpoint: area under the insulin concentration curve(AUCins) 0-6h | 0-6hour
  area under the insulin concentration curve
Pharmacokinetic endpoint: area under the insulin concentration curve(AUCins) 0-12h | 0-12hour
  area under the insulin concentration curve
Pharmacokinetic endpoint: area under the insulin concentration curve(AUCins)12-24h | 12-24hour
  area under the insulin concentration curve
Pharmacokinetic endpoint: area under the insulin concentration curve(AUCins).0-infinity | 0 to 24 hours
  area under the insulin concentration curve
Pharmacokinetic endpoint: time to maximum observed insulin concentration (tmax) | 0-24hour
  time to maximum observed insulin concentration
Pharmacokinetic endpoint: time(t)50%-ins(early) | 0-24hour
  time to half-maximum before Cins.max
Pharmacokinetic endpoint: time(t)50%-ins(late) | 0-24hour
  time to half-maximum after Cins.max
Pharmacokinetic endpoint: terminal elimination half-life (t½) | 0-24hour
  terminal elimination half-life calculated as t½=ln2/λz
Pharmacokinetic endpoint:terminal elimination rate constant(λz) | 0-24hour
  terminal elimination rate constant of insulin
Pharmacodynamic endpoints: area under the glucose infusion rate curve (AUCGIR) 0-2h | 0-2hour
  area under the glucose infusion rate curve
Pharmacodynamic endpoints: area under the glucose infusion rate curve (AUCGIR)0-6h | 0-6hour
  area under the glucose infusion rate curve
Pharmacodynamic endpoints: area under the glucose infusion rate curve(AUCGIR)0-12h | 0-12hour
  area under the glucose infusion rate curve
Pharmacodynamic endpoints: area under the glucose infusion rate curve (AUCGIR)12-24h | 12-24hour
  area under the glucose infusion rate curve
Pharmacodynamic endpoints: time to maximum glucose infusion rate (tGIR.max) | 0-24hour
  time to maximum glucose infusion rate
Pharmacodynamic endpoints: time to half-maximum glucose infusion rate before GIRmax(tGIR.50%-early) | 0-24hour
  time to half-maximum glucose infusion rate before Maximum glucose infusion rate(GIRmax)
Pharmacodynamic endpoints: time to half-maximum glucose infusion rate after GIRmax (tGIR.50%-late) | 0-24hour
  time to half-maximum glucose infusion rate after Maximum glucose infusion rate(GIRmax)
Pharmacodynamic endpoints: Onset of action | 0-24hour
  time from trial product administration until blood glucose concentration has decreased at least 5 mg/dL from baseline, where baseline is defined as the mean of blood glucose levels from -6, -4, and -2 minutes before trial product administration as measured by ClampArt(name of Clamp Devise).

OTHER OUTCOMES:
Safety endpoints: Number of subjects with Adverse Events, clinically significant changes in Physical examination, Vital signs. Local tolerability/ Injection site reactions | First dose to followup period (Total duration: 14 days approximate)
  Number of subjects with Adverse Events, clinically significant changes in Physical examination, Vital signs
  Local tolerability/ Injection site reactions
Safety endpoint: Number of subjects with clinically significant changes in Laboratory safety parameters, Electrocardiogram (ECG) | Screening and Follow-up period (Total duration: 35 days approximate)
  Number of subjects with clinically significant changes in Laboratory safety parameters.
  Number of subjects with clinically significant changes in Electrocardiogram (ECG)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Klein, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH Hellersbergstr. 9 D-41460 Neuss
Locations (2):
- Germany (2):
  - Profil Mainz GmbH & Co. KG Malakoff-Passage,Rheinstraße 4C D-55116, Mainz
  - Profil Institut für Stoffwechselforschung GmbH Hellersbergstr. 9 D-41460 Neuss, Neuss

IPD SHARING:
Plan to Share IPD: No